CLINICAL TRIAL: NCT07087028
Title: Comparison of Digital Anesthesia and Conventional Infiltration Techniques During Primary Tooth Extractions in Children
Brief Title: Digital vs. Conventional Anesthesia for Primary Tooth Extractions in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Özant Önçağ, Professsor, Ege University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16-3/7
Record Dates: First submitted 2024-10-09; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Pain Management; Dental Anxiety; Pediatric Dentistry; Dental Anesthesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FIRST Computerized Intraosseous Anesthesia (CCIA), SECOND Traditional Infiltration Anesthesia (TIA) (Experimental): In this randomized split-mouth crossover design, participants underwent two appointments for bilateral upper primary molar extractions. In this arm, at the first visit, computerized intraosseous anesthesia (CCIA) was administered using the SleeperOne™ system with a 30 G × 9 mm Effitec needle and 2% articaine with 1:100,000 epinephrine, followed by tooth extraction. At the second visit, conventional buccal infiltration anesthesia (TIA) was performed using a standard dental syringe and a 27-gauge needle on the contralateral molar, using the same anesthetic solution.
  Interventions: Device: SleeperOne™; Other: Conventional Infiltration Anesthesia
- FIRST Traditional Infiltration Anesthesia (TIA), SECOND (CCIA) (Experimental): In this randomized split-mouth crossover design, participants underwent two appointments for bilateral upper primary molar extractions. In this arm, at the first visit, conventional buccal infiltration anesthesia (TIA) was administered using a standard dental syringe and a 27-gauge needle, along with 2% articaine containing 1:100,000 epinephrine. At the second visit, computerized intraosseous anesthesia (CCIA) was delivered using the SleeperOne™ system with a 30 G × 9 mm Effitec needle, followed by extraction of the contralateral molar using the same anesthetic solution.
  Interventions: Device: SleeperOne™; Other: Conventional Infiltration Anesthesia

INTERVENTIONS:
Device: SleeperOne™ — Computerized intraosseous anesthesia was delivered using the SleeperOne™ (Dental HiTec, France) device with a 30 G × 9 mm Effitec needle at a 15° angle to the mucosa. A total of 2 mL 2% articaine with 1:100,000 epinephrine was administered per site.
Other: Conventional Infiltration Anesthesia — The intervention for the Conventional Infiltration Anesthesia involves the manual administration of a local anesthetic using a standard dental syringe with a fine-gauge needle.

SUMMARY:
This study aims to compare two different techniques of administering dental anesthesia to pediatric patients to determine which method causes less pain and anxiety during procedures like primary tooth extractions.

DETAILED DESCRIPTION:
Dental anxiety, particularly in pediatric patients, is a significant challenge, often triggered by fear of local anesthesia injections. Although local anesthesia aims to prevent pain during treatment, the injection process itself can cause anxiety and defensive behaviors, especially in children. To address this, various methods have been introduced to reduce discomfort, including topical anesthetics, slow injections, and thinner needles. However, traditional methods still face challenges in regulating injection rates, leading to the development of computer-controlled local anesthetic delivery (CCLAD) systems.

CCLAD, particularly intraosseous anesthesia systems like SleeperOne™, offer a controlled flow rate and pressure during anesthesia delivery, potentially reducing discomfort and anxiety. Despite numerous studies, results on the effectiveness of CCLAD in pediatric patients remain controversial. This study aims to bridge this gap by comparing the efficacy of computerized intraosseous anesthesia with conventional infiltration anesthesia in pediatric patients undergoing primary molar extraction. The goal is to assess pain perception and anxiety levels, with the hypothesis that intraosseous anesthesia may lead to better outcomes in terms of pain and anxiety reduction compared to conventional techniques.

The use of the SleeperOne™ device for intraosseous anesthesia is hypothesized to be more effective in reducing pain and anxiety compared to conventional infiltration techniques during the extraction of primary molars in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients in between 6-12 years old
* Physically and mentally healthy patients
* Cooperative patients who were rated as positive or definitely positive according to the Frankl behavior classification scale
* Patients who had primary molars that required extraction on both sides of maxillary arch.

Exclusion Criteria:

* Children allergic to local anesthetics
* Medically compromised and special children
* Teeth with hypoplasia
* Children who used analgesic drug 48 hours before treatment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Pain Perception - Visual Analogue Scale | During anesthesia and during extraction in each visit.
  Pain was assessed using a 10-centimeter Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse pain.
Pain Perception - Wong-Baker Faces Pain Rating Scale | During anesthesia and during extraction in each visit.
  Pain was assessed using the Wong-Baker Faces Pain Rating Scale (WBPRS), which ranges from 0 (no hurt) to 10 (hurts worst). Higher scores indicate worse pain.
Dental Anxiety - State-Trait Anxiety Inventory for Children - State Subscale | At baseline, after anesthesia and after extraction in each visit.
  Dental anxiety was assessed using the short form of the State-Trait Anxiety Inventory for Children - State Subscale (STAI-S). Scores range from 10 (low anxiety) to 40 (high anxiety).

SECONDARY OUTCOMES:
Physiological Arousal During Dental Procedure - Heart Rate | Before anesthesia, during anesthesia, and during extraction in each visit.
  Heart rate was measured using a pulse oximeter to monitor physiological arousal during the procedure. Heart rate may reflect a combination of pain, anxiety, and procedural stress. Unit of Measure is beats per minute (bpm). Higher values may indicate increased physiological arousal.
Baseline Dental Anxiety Assessed by Children's Fear Survey Schedule - Dental Subscale (CFSS-DS) | At the baseline before starting first visit.
  Baseline dental anxiety was assessed using the Children's Fear Survey Schedule - Dental Subscale (CFSS-DS), which includes 15 items scored from 1 to 5. Total scores range from 15 to 75. Higher scores indicate greater dental fear.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No